# STATISTICAL ANALYIS PLAN WITH RESULTS

Screen to Save: A Colorectal Cancer Educational Intervention

NCT03907579

Date: July 8, 2020

### ANALYSIS - BACKGROUND

For the Screen2Save intervention, subjects first take a survey, participate in the intervention and then take a final survey. The questions are the same on both surveys. All analysis was done using Stata/SE 15.1.

### DID THE INTERVENTION CHANGE THE SURVEY RESULTS?

We are most interested in whether the subjects scored better (had more correct answers) in the post survey than the pre survey. Thus, for analysis purposes, each question was coded as a dichotomous Correct or Not Correct. If a subject did not submit a response for the question, it was coded as Not Correct (we may want to revisit this).

In order to test whether there was a difference in the Correct responses in the pre and post tests, McNemar's Test was used.

The McNemar test is a non-parametric test for paired nominal data. It's used when you are interested in finding a change in proportion for the paired data. For example, you could use this test to analyze retrospective case-control studies, where each treatment is paired with a control. It could also be used to analyze an experiment where two treatments are given to matched pairs. This test is sometimes referred to as McNemar's Chi-Square test because the test statistic has a chi-square distribution. (https://www.statisticshowto.com/mcnemar-test/)

When sample sizes are small, the chi-squared value may not be well-approximated by the chi-squared distribution. The exact p-value can be computed.

Thus, for each pair of pre and post questions, McNemar's Test was performed and both the Chi<sup>2</sup> and the exact P-value are shown. If the p-value is significant (<0.05), then the null hypothesis (H0 = the number of correct responses on the pre survey are the same as on the post survey) can be rejected.

#### HOW DID THE SURVEY RESPONSE CHANGE?

Although the primary interest is whether the intervention increased knowledge about Colorectal cancer and screening, understanding what the specific responses were to the surveys is also of interest. CrossTab tables help to both quantify and visualize the relationship between the Pre and Post responses. The Pre responses are shown in the rows while the Post responses are in the columns. The light green to dark blue color gradient highlights the low to high number of responses for each category.

Did the intervention increase the number of correct answers?

In order to look at the overall impact of the intervention, the number of correct responses was tabulated for each participant pre and post intervention. This data is shown in a CrossTab table. As with the individual questions, no response/null answers were coded as incorrect. In order to test of the number of correct responses was significantly different pre and post intervention, the Wilcoxon Signed-Rank Test was used. This is the non-parametric (i.e. not normally distributed) equivalent of a paired t-test.

## SURVEY RESPONSES — WITH MCNEMAR'S CHI2 TEST STATISTIC AND EXACT P-VALUE AS WELL AS CROSSTAB

#### 1.COLORECTAL CANCER STARTS IN WHAT PART OF THE BODY?

Correct Answer: Colon and/or rectum

McNemar's chi2(1) = 0.00 Prob > chi2 = 1.0000 Exact McNemar significance probability = 1.0000

NOT SIGNIFICANT, THERE IS NOT A SIGNIFICANT DIFFERENCE IN THE CORRECT RESPONSES PRE AND POST SURVEY.

### Post Starts in what body part

| Pre Starts in what body part | Null | Colon and or rectum | Small<br>Intestine | Stomach | Grand Total |
|---|---|---|---|---|---|
| Null | 2 | 4 | 1 | | 7 |
| Colon and or rectum | 1 | 56 | 10 | 2 | 69 |
| Small Intestine | 1 | 8 | 10 | 1 | 20 |
| Stomach | | 1 | 1 | 2 | 4 |
| Grand Total | 4 | 69 | 22 | 5 | 100 |

### 2.A STOOL TEST (FIT/FOBT) CHECKS YOUR STOOL (POOP) FOR?

Correct Answer: Blood

McNemar's chi2(1) = 3.20 Prob > chi2 = 0.0736

Exact McNemar significance probability = 0.1153

| | Post Checks stool for | | | | | |
|---|---|---|---|---|---|---|
| Pre Checks<br>stool for | Null | Blood | Fat | Polyps | Tumors | Grand Total |
| Null | 3 | 6 | | 4 | 1 | 14 |
| Blood | 2 | 60 | 2 | 1 | 1 | 66 |
| Fat | | 2 | | | | 2 |
| Polyps | 1 | 5 | | 9 | 1 | 16 |
| Tumors | | 1 | | 1 | | 2 |
| Grand Total | 6 | 74 | 2 | 15 | 3 | 100 |

3. WHICH OF THE FOLLOWING ARE RISK FACTORS FOR COLORECTAL CANCER? PLEASE CHECK ALL THAT ARE CORRECT.

Correct Answer: Count of 5

McNemar's chi2(1) = 21.78 Prob > chi2 = 0.0000

Exact McNemar significance probability = 0.0000

| | Post Number of Risk Factors | | | | | |
|---|---|---|---|---|---|---|
| Pre Num | 1 | 2 | 3 | 4 | 5 | Grand Total |
| 0 | | 1 | | | 3 | 4 |
| 1 | 1 | 1 | | 3 | 8 | 13 |
| 2 | | 5 | 4 | 3 | 7 | 19 |
| 3 | 2 | | 2 | 1 | 6 | 11 |
| 4 | | | 1 | | 8 | 9 |
| 5 | | | 1 | 3 | 40 | 44 |
| Grand<br>Total | 3 | 7 | 8 | 10 | 72 | 100 |

### 4. IN GENERAL, A COLONOSCOPY SHOULD BE PERFORMED EVERY 10 YEARS STARTING AT AGE:

Correct Answer: 50

McNemar's chi2(1) = 13.00 Prob > chi2 = 0.0003

Exact McNemar significance probability = 0.0002



5. IN GENERAL, A STOOL (POOP) TEXT (FIT OR FOBT) SHOULD BE DONE EVERY YEAR STARTING AT AGE:

Correct Answer: 50

McNemar's chi2(1) = 20.16 Prob > chi2 = 0.0000

Exact McNemar significance probability = 0.0000

| | Post Stool test starting age | | | | | |
|---|---|---|---|---|---|---|
| Pre stool test<br>start age | Null | 30 | 40 | 50 | 60 | Grand Total |
| Null | 1 | | | 9 | | 10 |
| 30 | | 3 | 2 | 2 | | 7 |
| 40 | 1 | 1 | 8 | 7 | | 17 |
| 50 | | 1 | 2 | 44 | | 47 |
| 60 | | | 1 | 10 | 8 | 19 |
| Grand Total | 2 | 5 | 13 | 72 | 8 | 100 |

6. LYNCH SYNDROME IS A DISORDER THAT RUNS IN FAMILIES AND INCREASES MY CHANCES OF DEVELOPING COLORECTAL CANCER.

Correct Answer: True

McNemar's chi2(1) = 29.45 Prob > chi2 = 0.0000

Exact McNemar significance probability = 0.0000



7. THE EARLIER THAT COLORECTAL CANCER IS FOUND, THE GREATER MY CHANCES OF SURVIVAL.

Correct Answer: True

McNemar's chi2(1) = 2.00 Prob > chi2 = 0.1573

Exact McNemar significance probability = 0.5000



8. EVEN IF I HAVE NO SYMPTOMS, I MAY STILL HAVE COLORECTAL CANCER.

Correct Answer: True

McNemar's chi2(1) = 5.40 Prob > chi2 = 0.0201 Exact McNemar significance probability = 0.0352



 $9.\mathtt{POLYPS}$  ARE GROWTHS IN THE LINING OF THE COLON OR RECTUM THAT CAN DEVELOP INTO COLORECTAL CANCER.

Correct Answer: True

McNemar's chi2(1) = 0.00 Prob > chi2 = 1.0000

Exact McNemar significance probability = 1.0000

| Pre Poly | Post Polyps are growths<br>Null False True Grand Total | | | |
|---|---|---|---|---|
| Null | 1 | Tuise | 2 | 3 |
| True | 1 | 1 | 95 | 97 |
| Grand<br>Total | 2 | 1 | 97 | 100 |

10. A COLONOSCOPY CAN BE USED TO FIND POLYPS IN THE COLON AND RECTUM.

Correct Answer: True

McNemar's chi2(1) = 1.00 Prob > chi2 = 0.3173

Exact McNemar significance probability = 1.0000



11. A DIET HIGH IN RED MEATS AND PROCESSED MEATS (LUNCH MEATS, HOT DOGS) INCREASES MY CHANCES OF DEVELOPING COLORECTAL CANCER.

Correct Answer: True

McNemar's chi2(1) = 3.00 Prob > chi2 = 0.0833

Exact McNemar significance probability = 0.1460



### 12. IT IS OK TO SKIP COLORECTAL CANCER SCREENING IF I DO NOT HAVE ANY SYMPTOMS.

Correct Answer: False

McNemar's chi2(1) = 0.33 Prob > chi2 = 0.5637

Exact McNemar significance probability = 0.7744

| | Post Skip Screening | | | |
|----------------|---------------------|-------|------|-------------|
| Pre Skip | Null | False | True | Grand Total |
| Null | 1 | 2 | | 3 |
| False | | 87 | 7 | 94 |
| True | | 3 | | 3 |
| Grand<br>Total | 1 | 92 | 7 | 100 |

### 13. MY CHANCES OF DEVELOPING COLORECTAL CANCER ARE HIGHER IF SOMEONE IN MY IMMEDIATE FAMILY HAS IT OR HAS HAD IT.

Correct Answer: True

McNemar's chi2(1) = 4.50 Prob > chi2 = 0.0339

Exact McNemar significance probability = 0.0703

Chi2 is significant, but Exact p-value is not significant. Since the Incorrect responses (when added together) have a cellsize <4, then the Exact P-value should be used.



### 14. INCREASING MY PHYSICAL ACTIVITY WILL NOT LOWER MY CHANCES OF DEVELOPING COLORECTAL CANCER.

Correct Answer: False

McNemar's chi2(1) = 5.83 Prob > chi2 = 0.0158

Exact McNemar significance probability = 0.0241



### TOTAL NUMBER OF CORRECT ANSWERS

| | | | Pos | t Total Cor | rect Answ | ers | | |
|-----------|---|---|-----|-------------|-----------|-----|-----|---------|
| Pre Total | 8 | 9 | 10 | 11 | 12 | 13 | Yes | Grand T |
| 4 | | 1 | | | | | | 1 |
| 6 | | | 1 | 1 | | | | 2 |
| 7 | 1 | | 1 | | | 1 | | 3 |
| 8 | 1 | 1 | | 2 | 1 | 1 | | 6 |
| 9 | | | 2 | | 4 | | | 6 |
| 10 | 2 | 2 | 4 | 7 | 3 | 4 | | 22 |
| 11 | | | 2 | | 8 | 6 | | 16 |
| 12 | | | | 5 | 9 | 10 | | 24 |
| 13 | | | | 2 | 5 | 5 | | 12 |
| 14 | | | 1 | | 1 | 5 | | 7 |
| Yes | | | | | | | 1 | 1 |
| Grand To | 4 | 4 | 11 | 17 | 31 | 32 | 1 | 100 |

### Wilcoxon Signed Rank Test

| Sign | Obs | Sum ranks | Expected |
|----------|-----|-----------|----------|
| Positive | 25 | 1318 | 2420 |
| Negative | 55 | 3522 | 2420 |
| Zero | 20 | 210 | 210 |
| All | 100 | 5050 | 5050 |

unadjusted variance 84587.50 adjustment for ties -2388.38 adjustment for zeros -717.50

\_\_\_\_\_

adjusted variance 81481.63

Ho: preTotalCorrect = postTotalCorrect

z = -3.861

Prob > |z| = 0.0001

### SUMMARY STATISTICS

### **Pre Total Correct Answers**

| | Percentiles | Smallest | | |
|-----|-------------|----------|-------------|-----------|
| 1% | 2.5 | 1 | | |
| 5% | 7 | 4 | | |
| 10% | 8 | 6 | Obs | 100 |
| 25% | 10 | 6 | Sum of Wgt. | 100 |
| 50% | 11 | | Mean | 10.78 |
| | | Largest | Std. Dev. | 2.195404 |
| 75% | 12 | 14 | | |
| 90% | 13 | 14 | Variance | 4.819798 |
| 95% | 14 | 14 | Skewness | -1.335507 |
| 99% | 14 | 14 | Kurtosis | 6.343168 |

### **Post Total Correct Answers**

| | Percentiles | Smallest | | |
|-----|-------------|----------|-------------|-----------|
| 1% | 4.5 | 1 | | |
| 5% | 8.5 | 8 | | |
| 10% | 10 | 8 | Obs | 100 |
| 25% | 11 | 8 | Sum of Wgt. | 100 |
| 50% | 12 | | Mean | 11.54 |
| | | Largest | Std. Dev. | 1.719878 |
| 75% | 13 | 13 | | |
| 90% | 13 | 13 | Variance | 2.95798 |
| 95% | 13 | 13 | Skewness | -2.702217 |
| 99% | 13 | 13 | Kurtosis | 15.56301 |

| Variable | Obs | Mean | Std. Dev. | Min | Max |
|------------------|-----|-------|-----------|-----|-----|
| preTotalCorrect | 100 | 10.78 | 2.195404 | 1 | 14 |
| postTotalCorrect | 100 | 11.54 | 1.719878 | 1 | 13 |

The 1<sup>st</sup> column is Total Correct Answers Post – Pre. So, one person (Freq column) had 4 more correct answers on the pre test and one person had 6 more correct answers Post. In most cases (29), people had one more correct answer.

| Post – Pre Total Correct | Freq. | Percent | Cum. |
|--------------------------|-------|---------|--------|
| -4 | 1 | 1.00 | 1.00 |
| -2 | 5 | 5.00 | 6.00 |
| -1 | 19 | 19.00 | 25.00 |
| 0 | 20 | 20.00 | 45.00 |
| 1 | 29 | 29.00 | 74.00 |
| 2 | 9 | 9.00 | 83.00 |
| 3 | 11 | 11.00 | 94.00 |
| 4 | 2 | 2.00 | 96.00 |
| 5 | 3 | 3.00 | 99.00 |
| 6 | 1 | 1.00 | 100.00 |
| Total | 100 | 100.00 | |

### INTENT

No analysis was done on the intent questions as they were only asked one time.

### Intent

